CLINICAL TRIAL: NCT05117723
Title: Intraductal Papillary Mucinous Neoplasm (IPMN) Database - A Tool to Predict Pancreatic Cancer
Acronym: MAPS
Status: Recruiting | Type: Observational
Sponsor: St Vincent's Hospital Melbourne (Other)
Collaborators: Epworth Healthcare (Other)
Responsible Party: Principal Investigator, Adrian Fox, Principal Investigator, St Vincent's Hospital Melbourne
Other Study IDs: 76739
Record Dates: First submitted 2021-10-21; First posted 2021-11-11 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: IPMN, Pancreatic; IPMN
Keywords: pancreatic cyst
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cancer is the 5th leading cause of cancer death in Australia. Surgery remains the most effective treatment for early pancreatic cancer and currently the only potential for cure. Unfortunately, many patients present with advanced disease and are not suitable for surgery. Therefore, it is vital to detect these cancers early. In the absence of significant data from prospective studies, all of the guidelines are based on a critical review of available data and consensus of experts. The primary aim is to delineate the progression of IPMN to pancreatic malignancy as confirmed by surgical pathology, radiology and biochemical diagnosis. The secondary aims are (i) To outline the management of IPMNs for those who have progressed straight to surgery or surveillance by endoscopic ultrasound (EUS) (ii)To validate the International consensus guidelines for management of IPMN - Fukuoka consensus guidelines and tertiary aim to identify potential risk factors, if any that increase risk of malignancy within the IPMNs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the age of 18 and 90 years old who have been identified with a cystic mass consistent with IPMN on imaging

Exclusion Criteria:

* Patients who formally decline enrolment into the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with IPMN will be identified from consultations at each hospital site with surgical and medical specialists with an interest in pancreatic conditions. This will occur via consultations conducted in public clinic settings and from private consultations and multi-disciplinary meetings.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-26 (Actual); Primary Completion 2031-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients who have progressed to further investigations including endoscopic ultrasound (EUS) and/or surgical intervention. | From diagnosis of IPMN followed by clinical follow ups at 3, 6 or 12 monthly interval as specified by clinician, up to 10 years
Risk stratification for patients with IPMN into those that require more intensive screening and possibly intervention versus those that are unlikely to progress to malignancy. | From diagnosis of IPMN followed by clinical follow ups at 3, 6 or 12 monthly interval as specified by clinician, up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Fox, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital Melbourne, Fitzroy, Victoria, Australia